CLINICAL TRIAL: NCT01091246
Title: A Randomized, Double-Blind, Active Controlled Study to Evaluate the Immunogenicity of Quadrivalent LAIV in Children
Brief Title: A Study to Evaluate the Immunogenicity of Quadrivalent Live Attenuated Influenza Vaccine (LAIV) in Children
Acronym: LAIV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Judith Falloon, M.D., MedImmune, LLC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MI-CP208
Record Dates: First submitted 2010-03-19; First posted 2010-03-23 (Estimated); Results first posted 2011-09-22 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: Healthy or Stable Chronic Illness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Q/LAIV (MEDI3250) (Experimental): Q/LAIV (quadrivalent live attenuated influenza vaccine) (MEDI3250) was supplied in the Becton Dickinson Accuspray device that delivers a 0.2 mL total volume intranasal dose divided into each nostril (ie, administered as 0.1 mL per nostril). Each 0.2 mL dose contained 10^7.0 ± 0.5 fluorescent focus units (FFU) of each of 4 temperature sensitive, cold-adapted, attenuated, 6:2 resassortant influenza strains (A/H1N1 [A/South Dakota/6/2007], A/H3N2 [A/Uruguay/716/2007], B/Victoria [B/Malaysia/2506/2004], and B/Yamagata [B/Florida/4/2006]).
  Interventions: Biological: Q/LAIV (MEDI3250)
- FluMist/B/Yamagata (Experimental): FluMist/B/Yamagata (trivalent live attenuated influenza vaccine) was supplied in the BD Accuspray device that delivers a 0.2 mL total volume intranasal dose divided into each nostril (ie, administered as 0.1 mL per nostril). Each 0.2 mL dose contained 10^7.0 ± 0.5 FFU of each of 3 temperature sensitive, cold-adapted, attenuated, 6:2 reassortant influenza strains (A/H1N1 [South Dakota/6/2007], A/H3N2 [A/Uruguay/716/2007], and B/Yamagata [B/Florida/4/2006])
  Interventions: Biological: FluMist/B/Yamagata
- FluMist/B/Victoria (Experimental): FluMist/B/Victoria (trivalent live attenuated influenza vaccine) was supplied in the BD Accuspray device that delivers a 0.2 mL total volume intranasal dose divided into each nostril (ie, administered as 0.1 mL per nostril). Each 0.2 mL dose contained 10^7.0 ± 0.5 FFU of each of 3 temperature sensitive, cold-adapted, attenuated, 6:2 reassortant influenza stains (A/H1N1 [A/South Dakota/6/2007], A/H3N2 [A/Uruguay/716/2007], and B/Victoria [B/Malaysia/2506/2004]).
  Interventions: Biological: FluMist/B/Victoria

INTERVENTIONS:
Biological: Q/LAIV (MEDI3250) — 10 ^7.0 ± 0.5 FFU/dose of each of 4 influenza virus strains: A/H1N1, A/H3N2, B/Yamagata, and B/Victoria
  Arms: Q/LAIV (MEDI3250)
Biological: FluMist/B/Yamagata — 10 ^7.0 ± 0.5 FFU/dose of each of 3 influenza virus strains: A/H1N1, A/H3N2, and B/Yamagata
  Arms: FluMist/B/Yamagata
Biological: FluMist/B/Victoria — 10 ^7.0 ± 0.5 FFU/dose of each of 3 influenza virus strains: A/H1N1, A/H3N2, and B/Victoria
  Arms: FluMist/B/Victoria

SUMMARY:
The primary objective of this study is to demonstrate the immunologic noninferiority of Q/LAIV to FluMist in children 2 to 17 years of age.

DETAILED DESCRIPTION:
The randomized, double-blind study was designed to demonstrate the immunologic noninferiority of Q/LAIV compared to FluMist in children 2-17 years by comparing the strain-specific post-dose geometric mean titers of hemagglutination inhibition antibodies. Children were randomized 3:1:1 to receive Q/LAIV or one of two FluMist vaccines. Subjects 9-17 years of age received a single dose, and those 2-8 years of age received two doses one month apart. Serum was obtained 1 month after dose 1 except in influenza vaccine-naive subjects 2-8 years old, when it was obtained after dose 2. Safety and tolerability were also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 2 through 17 years at the time of randomization
* Written informed consent and any locally required authorization (eg, HIPAA in the USA, EU Data Privacy Directive in the EU, and written informed assent if applicable) obtained from the subject/legal representative prior to performing any protocol-related procedures, including screening evaluations
* Females of childbearing potential, unless surgically sterile (ie, bilateral tubal ligation, bilateral oophorectomy, or hysterectomy), has sterile male partner, is premenarchal, or practices abstinence, must have used an effective method of avoiding pregnancy (including oral, transdermal, or implanted contraceptives, intrauterine device, female condom with spermicide, diaphragm with spermicide, cervical cap with spermicide, or use of a condom with spermicide by the sexual partner) for 30 days prior to the first dose of investigational product, and must agree to continue using such precautions for 60 days after the final dose of investigational product
* A subject who is considered by the investigator to be at risk of pregnancy must also have a negative urine pregnancy test at screening and, if screening and Day 0 do not occur on the same day, on the day of vaccination prior to randomization. Investigator judgment is required to assess each subject's need for pregnancy testing
* Healthy by medical history and physical examination OR presence of stable underlying chronic medical condition for which hospitalization has not been required in the previous year
* Able to complete follow-up period of 180 days post last dose of vaccine as required by the protocol
* Subject/legal representative is available by telephone
* Child's legal representative is able to understand and comply with the requirements of the protocol, as judged by the investigator

Exclusion Criteria:

* Acute illness or evidence of significant active infection at randomization;
* Fever ≥ 100.4°F (38.0°C) at randomization
* History of asthma, or in children < 5 years of age, history of recurrent wheezing
* Any drug therapy from 15 days prior to randomization or expected drug therapy through 28 days post last dose with the exception of the following classes/types of medications, which are allowed:
* Contraceptives (change in contraceptive type or method is acceptable as long as guidelines are followed for prevention of pregnancy during change);
* Topical corticosteroids, calcineurin inhibitors, or antifungals for uncomplicated dermatitis;
* Chronic medications (including those taken on an as-needed basis) that have been well tolerated and were not initiated and/or did not have a dosage change within 90 days prior to randomization.
* Current or expected receipt of immunosuppressive medications within a 28 day window around any dose, including an immunosuppressive dose of corticosteroids, which is defined as ≥ 20 mg/day of prednisone or its equivalent, given daily or on alternate days for ≥ 15 days) (intranasal, intra-articular, and topical corticosteroids are permitted); Note: topical corticosteroids for uncomplicated dermatitis may be used throughout the study according to the judgment of the investigator; topical calcineurin inhibitors may be used in accordance with their package insert at entry and during study participation
* Receipt of immunoglobulin or blood products within 90 days before randomization into the study or expected receipt during study participation
* Receipt of any investigational drug therapy within 28 days prior to Dose 1 or planned receipt of any investigational drug therapy through 90 days after final dosing of investigational product (use of licensed agents for indications not listed in the package insert is permitted)
* Receipt of any nonstudy vaccine within 28 days prior to randomization or planned receipt of nonstudy vaccine through 28 days after final dosing
* Receipt of any nonstudy seasonal influenza vaccine within 90 days of Dose 1 or planned receipt of nonstudy seasonal influenza vaccine prior to 35 days post last dose of investigational product
* Any known immunosuppressive condition or immune deficiency disease including known or suspected infection with human immunodeficiency virus (HIV)
* History of allergic disease or reactions likely to be exacerbated by any component of the investigational product including allergy to eggs, egg proteins, gentamicin, or gelatin or serious, life threatening, or severe reactions to previous influenza vaccinations
* Use of aspirin or salicylate-containing products within 28 days prior to randomization or expected receipt through 28 days after final vaccination;
* History of Guillain-Barré syndrome
* Use of antiviral agents with activity against influenza virus (including amantadine, rimantadine, oseltamivir, and zanamivir) within 28 days prior to first dose of investigational product or anticipated use of such agents within 28 days after last scheduled vaccination
* Known or suspected mitochondrial encephalomyopathy
* Pregnant or lactating female
* History of alcohol or drug abuse that, in the opinion of the investigator, would affect the subject's safety or compliance with study
* Any condition that, in the opinion of the investigator, might compromise the safety of the subject in the study or would interfere with evaluation of the safety or immunogenicity of the investigational products
* Subject, legal representative, or immediate family member of subject who is an employee of the clinical study site or who is otherwise involved with the conduct of the study
* A history of epilepsy, seizure, or an evolving neurological condition except that of a single febrile seizure that occurred 3 or more years prior to enrollment would not disqualify a subject

Note: an individual who initially is excluded from study participation based on one or more of the above time-limited criteria may be reconsidered for enrollment once the condition has resolved as long as the subject continues to meet all other entry criteria and the same SID number is used

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2312 (Actual)
Dates: Start 2010-03; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Falloon, M.D., Study Director — MedImmune LLC
Locations (98):
- United States (98):
  - Research Site, Birmingham, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Tucson, Arizona
  - Research Site, Benton, Arkansas
  - Research Site, Bentonville, Arkansas
  - Research Site, Fayetteville, Arkansas
  - Research Site, Jonesboro, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Fountain Valley, California
  - Research Site, Fresno, California
  - Research Site, Long Beach, California
  - Research Site, Paramount, California
  - Research Site, Sacramento, California
  - Research Site, San Francisco, California
  - Research Site, West Covina, California
  - Research Site, Wilmington, Delaware
  - Research Site, Boca Raton, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Ponte Vedra, Florida
  - Research Site, South Miami, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Dalton, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Woodstock, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, DeKalb, Illinois
  - Research Site, Newton, Kansas
  - Research Site, Overland Park, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Bardstown, Kentucky
  - Research Site, Lexington, Kentucky
  - Research Site, Metairie, Louisiana
  - Research Site, Kalamazoo, Michigan
  - Research Site, Niles, Michigan
  - Research Site, Stevensville, Michigan
  - Research Site, Plymouth, Minnesota
  - Research Site, Saint Paul, Minnesota
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Papillion, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Lebanon, New Hampshire
  - Research Site, Albuquerque, New Mexico
  - Research Site, Binghamton, New York
  - Research Site, Brooklyn, New York
  - Research Site, Mineola, New York
  - Research Site, Rochester, New York
  - Research Site, Asheboro, North Carolina
  - Research Site, Boone, North Carolina
  - Research Site, Clyde, North Carolina
  - Research Site, Mt Pleasant, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Bismarck, North Dakota
  - Research Site, Fargo, North Dakota
  - Research Site, Akron, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Huber Heights, Ohio
  - Research Site, Norman, Oklahoma
  - Research Site, Yukon, Oklahoma
  - Research Site, Altoona, Pennsylvania
  - Research Site, Erie, Pennsylvania
  - Research Site, Greenville, Pennsylvania
  - Research Site, Harleysville, Pennsylvania
  - Research Site, Hermitage, Pennsylvania
  - Research Site, Latrobe, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Scotland, Pennsylvania
  - Research Site, Sellersville, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Bristol, Tennessee
  - Research Site, Clarksville, Tennessee
  - Research Site, Kingsport, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Longview, Texas
  - Research Site, New Branfels, Texas
  - Research Site, Sugarland, Texas
  - Research Site, Draper, Utah
  - Research Site, Layton, Utah
  - Research Site, Orem, Utah
  - Research Site, Roy, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, South Jordan, Utah
  - Research Site, Syracuse, Utah
  - Research Site, Burke, Virginia
  - Research Site, Charlottesville, Virginia
  - Research Site, Vienna, Virginia
  - Research Site, Virginia Beach, Virginia
  - Research Site, Huntington, West Virginia
  - Research Site, Franklin, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 2,481 participants provided written informed consent and were screened for the study. Of these, 2,312 participants were randomized into the study between 29Mar2010 to 12May2010 at 97 sites in the USA.
Pre-assignment Details: Eligible participants were randomized in a 3:1:1 ratio to receive Q/LAIV, FluMist/B/Yamagata, or FluMist/B/Victoria. Randomization was stratified by age (2 to 8 years, 9 to 17 years). For subjects 2 to 8 years of age only, randomization was also stratified by previous seasonal influenza vaccination history.
Groups:
- Q/LAIV (MEDI3250): Q/LAIV (quadrivalent live attenuated influenza vaccine) (MEDI3250) was supplied in the Becton Dickinson (BD) Accuspray device that delivers a 0.2 mL total volume intranasal dose divided into each nostril (ie, administered as 0.1 mL per nostril). Each 0.2 mL dose contained 10^7.0 ± 0.5 fluorescent focus units (FFU) of each of 4 temperature sensitive, cold-adapted, attenuated, 6:2 resassortant influenza strains (A/H1N1 [A/South Dakota/6/2007], A/H3N2 [A/Uruguay/716/2007], B/Victoria [B/Malaysia/2506/2004], and B/Yamagata [B/Florida/4/2006]).
Period: Overall Study
Arm/Group | Q/LAIV (MEDI3250) | FluMist/B/Yamagata | FluMist/B/Victoria
Started | 1385 | 464 | 463
Completed | 1350 | 448 | 450
Not Completed | 35 | 16 | 13
Not completed — Lost to Follow-up | 23 | 11 | 7
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Withdrawal by Subject | 9 | 5 | 4
Not completed — Subject not dosed | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Q/LAIV (MEDI3250) | FluMist/B/Yamagata | FluMist/B/Victoria | Total
Number analyzed (Participants) | 1385 | 464 | 463 | 2312
Age Continuous [Mean (Standard Deviation); unit: Years] | 6.7 (3.8) | 6.8 (3.8) | 6.8 (3.9) | 6.7 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 707 | 229 | 240 | 1176
  Male | 678 | 235 | 223 | 1136

OUTCOME MEASURES:

1. Primary Outcome: The 4 Post-dose Strain-specific Serum Hemagglutination Inhibition (HAI) Antibody Geometric Mean Titers (GMT) in the Q/LAIV (MEDI3250) Arm Are Noninferior to Those in the Comparator FluMist Group.
Description: Noninferior immune response was defined as having the upper bound of the 2-sided 95% confidence intervals (CIs) for the HAI antibody GMT ratio (FluMist comparator divided by Q/LAIV) ≤ 1.5 for each of the 4 strains. .
Time Frame: Day 28 post immunogenicity dose
Population: All participants who received any investigational product (Q=1385; FY=464; FV=463; All FM=927), had post dose HAI antibody measurement at the appropriate time and had no protocol deviation judged to have the potential to interfere with the generation or interpretation of an immune response (Q=1327; FY=445; FV=437; All FM=883).
Measure: Geometric Mean (Full Range); unit: Geometric mean titer
Groups:
- All FluMist Group: All FluMist group for A/H1N1 and A/H3N2 strains, where data from both the FluMist/B/Yamagata arm and the FluMist/B/Victoria arm were combined
Arm/Group | Q/LAIV (MEDI3250) | FluMist/B/Yamagata | FluMist/B/Victoria | All FluMist Group
Number analyzed (Participants) | 1327 | 445 | 437 | 883
Geometric mean titer
  A/H1N1 | 16.7 [15.9 to 17.6] | NA [NA to NA] — The comparators for the GMT ratios for the primary endpoint were participants in the All FluMist group (combined data for both FluMist arms) for A/H1N1 and A/H3N2 strains. | NA [NA to NA] — The comparators for the GMT ratios for the primary endpoint were participants in the All FluMist group (combined data for both FluMist arms) for A/H1N1 and A/H3N2 strains. | 17.9 [16.8 to 19.1]
  A/H3N2 | 27.7 [26.1 to 29.4] | NA [NA to NA] — The comparators for the GMT ratios for the primary endpoint were participants in the All FluMist group (combined data for both FluMist arms) for A/H1N1 and A/H3N2 strains. | NA [NA to NA] — The comparators for the GMT ratios for the primary endpoint were participants in the All FluMist group (combined data for both FluMist arms) for A/H1N1 and A/H3N2 strains. | 28.8 [26.7 to 31.1]
  B/Yamagata | 49.6 [46.6 to 52.8] | 59.8 [53.7 to 66.7] | NA [NA to NA] — B/Yamagata strain not in the investigational product. | NA [NA to NA] — The comparators for the GMT ratios for the primary endpoint were participants in the All FluMist group (combined data for both FluMist arms) for A/H1N1 and A/H3N2 strains.
  B/Victoria | 35.4 [33.3 to 37.7] | NA [NA to NA] — B/Victoria strain not in the investigational product. | 37.0 [33.4 to 41.0] | NA [NA to NA] — The comparators for the GMT ratios for the primary endpoint were participants in the All FluMist group (combined data for both FluMist arms) for A/H1N1 and A/H3N2 strains.
Statistical Analysis 1: Comparison: Q/LAIV (MEDI3250) vs All FluMist Group; A/H1N1: The statistical hypothesis testing for the primary endpoint for Q/LAIV was: H0: Rj > 1.5, for any j HA: Rj ≤ 1.5, for all j Where Rj was any of the 4 strain-specific post immunogenicity dose GMT ratios: (FluMist/B/Yamagata + FluMist/B/Victoria) / (Q/LAIV) for A/H1N1 strain; Test type: Non-Inferiority or Equivalence — The noninferior immune response was assessed by evaluating the upper bound of the two-sided 95% confidence intervals for the strain specific HAI antibody GMT ratios (FluMist divided by Q/LAIV) to the noninferiority margin of 1.5; Bootstrapping; Ratio of geometric mean = 1.07, 95% CI 2-sided [0.98 to 1.16]
Statistical Analysis 2: Comparison: Q/LAIV (MEDI3250) vs All FluMist Group; A/H3N2: The statistical hypothesis testing for the primary endpoint for Q/LAIV was: H0: Rj > 1.5, for any j HA: Rj ≤ 1.5, for all j Where Rj was any of the 4 strain-specific post immunogenicity dose GMT ratios: (FluMist/B/Yamagata + FluMist/B/Victoria) / (Q/LAIV) for A/H3N2 strain; Test type: Non-Inferiority or Equivalence — The noninferior immune response was assessed by evaluating the upper bound of the two-sided 95% confidence intervals for the strain specific HAI antibody GMT ratios (FluMist divided by Q/LAIV) to the noninferiority margin of 1.5. If the upper bounds of 95% CIs were ≤ 1.5 for all 4 strains, the immunologic noninferiority of Q/LAIV compared to FluMist was declared; Bootstrapping; Ratio of geometric means = 1.04, 95% CI 2-sided [0.94 to 1.14]
Statistical Analysis 3: Comparison: Q/LAIV (MEDI3250) vs FluMist/B/Yamagata; B/Yamagata: The statistical hypothesis testing for the primary endpoint for Q/LAIV was: H0: Rj > 1.5, for any j HA: Rj ≤ 1.5, for all j Where Rj was any of the 4 strain-specific post immunogenicity dose GMT ratios: (FluMist/B/Yamagata) / (Q/LAIV) for B/Yamagata strain; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Ratio of geometric mean = 1.21, 95% CI 2-sided [1.07 to 1.37]
Statistical Analysis 4: Comparison: Q/LAIV (MEDI3250) vs FluMist/B/Victoria; B/Victoria: The statistical hypothesis testing for the primary endpoint for Q/LAIV was: H0: Rj > 1.5, for any j HA: Rj ≤ 1.5, for all j Where Rj was any of the 4 strain-specific post immunogenicity dose GMT ratios: (FluMist/B/Victoria) / (Q/LAIV) for B/Victoria strain; Test type: Non-Inferiority or Equivalence — The noninferior immune response was assessed by evaluating the upper bound of the two-sided 95% confidence intervals for the strain specific HAI antibody GMT ratios (FluMist divided by Q/LAIV) to the noninferiority margin of 1.5. If the upper bounds of 95% confidence intervals were ≤ 1.5 for all 4 strains, the immunologic noninferiority of Q/LAIV compared to FluMist was declared; Ratio of geometric mean = 1.05, 95% CI 2-sided [0.93 to 1.18]

2. Secondary Outcome: The Percent of Participants (Regardless of Serostatus) Within Each Treatment Arm Who Experienced a Seroresponse to the A/H1N1 Strain Post Immunogenicity Dose
Description: Seroresponse was defined as a ≥ 4-fold rise in HAI antibody titer from baseline.
Time Frame: Day 0 and Day 28 post immunogenicity dose
Population: All participants who received any investigational product (Q=1385; All FM=927), had post dose HAI antibody measurement at the appropriate time, and had no protocol deviation judged to have the potential to interfere with the generation or interpretation of an immune response (Q=1320; All FM=878).
Measure: Number; unit: percent of participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist Group
Number analyzed (Participants) | 1320 | 878
percent of participants | 6.3 | 8.2

3. Secondary Outcome: Percent of Participants (Regardless of Serostatus) Within Each Treatment Arm Who Experienced a Seroresponse to the A/H3N2 Strain Post Immunogenicity Dose
Description: Seroresponse was defined as a ≥ 4-fold rise in HAI antibody titer from baseline.
Time Frame: Day 0 and Day 28 post immunogenicity dose
Population: All participants who received any investigational product (Q=1385; All FM=927), had post dose HAI antibody measurement at the appropriate time and had no protocol deviation judged to have the potential to interfere with the generation or interpretation of an immune response (Q=1321; All FM=879).
Measure: Number; unit: Percent of participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist Group
Number analyzed (Participants) | 1321 | 879
Percent of participants | 3.9 | 3.6

4. Secondary Outcome: Percent of Participants (Regardless of Serostatus) Within Each Treatment Arm Who Experienced a Seroresponse to the B/Yamagata Strain Post Immunogenicity Dose
Description: Seroresponse was defined as a ≥ 4-fold rise in HAI antibody titer from baseline.
Time Frame: Day 0 and Day 28 post immunogenicity dose
Population: All participants who received any investigational product (Q=1385; FY=464), had post dose HAI antibody measurement at the appropriate time, and had no protocol deviation judged to have the potential to interfere with the generation or interpretation of an immune response (Q=1321; FY=441).
Measure: Number; unit: Percent of participants
Arm/Group | Q/LAIV (MEDI3250) | FluMist/B/Yamagata
Number analyzed (Participants) | 1321 | 441
Percent of participants | 43.4 | 44.9

5. Secondary Outcome: Percent of Participants (Regardless of Serostatus) Within Each Treatment Arm Who Experienced a Seroresponse to the B/Victoria Strain Post Immunogenicity Dose
Description: Seroresponse was defined as a ≥ 4-fold rise from baseline.
Time Frame: Day 0 and Day 28 post immunogenicity dose
Population: All participants who received any investigational product (Q=1385; FV=463), had post dose HAI antibody measurement at the appropriate time, and had no protocol deviation judged to have the potential to interfere with the generation or interpretation of an immune response (Q=1321; FV=437).
Measure: Number; unit: Percent of participants
Arm/Group | Q/LAIV (MEDI3250) | FluMist/B/Victoria
Number analyzed (Participants) | 1321 | 437
Percent of participants | 39.1 | 38.4

6. Secondary Outcome: Percent of Serosusceptible Participants Within Each Treatment Arm Who Experienced a Seroresponse to the A/H1N1 Strain Post Immunogenicity Dose
Description: Serosusceptible was defined as a baseline HAI titer ≤ 8. Seroresponse was defined as a ≥ 4-fold rise in HAI titer from baseline.
Time Frame: Day 0 and Day 28 post immunogenicity dose
Population: All participants who received any investigational product (Q=1385; All FM=927), had post dose HAI antibody measurement at the appropriate time, had no protocol deviation judged to have the potential to interfere with the generation or interpretation of an immune response, and were serosusceptible to the strain (Q=569; All FM=392).
Measure: Number; unit: Percent of participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist Group
Number analyzed (Participants) | 569 | 392
Percent of participants | 12.7 | 17.6

7. Secondary Outcome: Percent of Serosusceptible Participants Within Each Treatment Arm Who Experience Seroresponse to the A/H3N2 Strain Post Immunogenicity Dose
Description: as for outcome 6
Time Frame: Day 0 and Day 28 post immunogenicity dose
Population: All participants who received any investigational product (Q=1385; All FM=927), had post dose HAI antibody measurement at the appropriate time, had no protocol deviation judged to have the potential to interfere with the generation or interpretation of an immune response, and were serosusceptible to the strain (Q=435; All FM=298).
Measure: Number; unit: Percent of participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist Group
Number analyzed (Participants) | 435 | 298
Percent of participants | 9.9 | 9.4

8. Secondary Outcome: Percent of Serosusceptible Participants Within Each Treatment Arm Who Experience Seroresponse to the B/Yamagata Strain Post Immunogenicity Dose
Description: as for outcome 6
Time Frame: Day 0 and Day 28 post immunogenicity dose
Population: All participants who received any investigational product (Q=1385; FY=464), had post dose HAI antibody measurement at the appropriate time, had no protocol deviation judged to have the potential to interfere with the generation or interpretation of an immune response, and were serosusceptible to the strain (Q=588; FY=192).
Measure: Number; unit: Percent of participants
Arm/Group | Q/LAIV (MEDI3250) | FluMist/B/Yamagata
Number analyzed (Participants) | 588 | 192
Percent of participants | 79.1 | 81.3

9. Secondary Outcome: Percent of Serosusceptible Participants Within Each Treatment Arm Who Experience Seroresponse to the B/Victoria Strain Post Immunogenicity Dose
Description: as for outcome 6
Time Frame: Day 0 and Day 28 post immunogenicity dose
Population: All participants who received any investigational product (Q=1385; FV=463), had post dose HAI antibody measurement at the appropriate time, had no protocol deviation judged to have the potential to interfere with the generation or interpretation of an immune response, and were serosusceptible to the strain (Q=620; FV=191).
Measure: Number; unit: Percent of participants
Arm/Group | Q/LAIV (MEDI3250) | FluMist/B/Victoria
Number analyzed (Participants) | 620 | 191
Percent of participants | 66.1 | 69.6

10. Secondary Outcome: Percent of Seronegative Participants Within Each Treatment Arm Who Experienced a Seroresponse to the A/H1N1 Strain Post Immunogenicity Dose
Description: Seronegative was defined as a baseline HAI titer ≤ 4. Seroresponse was defined as a ≥ 4-fold rise in HAI titer from baseline.
Time Frame: Day 0 and Day 28 post immunogenicity dose
Population: All participants who received any investigational product (Q=1385; All FM=927), had post dose HAI antibody measurement at the appropriate time, and had no protocol deviation judged to have the potential to interfere with the generation or interpretation of an immune response and were seronegative to the strain (Q=460; All FM=321).
Measure: Number; unit: Percent of participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist Group
Number analyzed (Participants) | 460 | 321
Percent of participants | 14.6 | 19.6

11. Secondary Outcome: Percent of Seronegative Participants Within Each Treatment Arm Who Experienced a Seroresponse to the A/H3N2 Strain Post Immunogenicity Dose
Description: as for outcome 10
Time Frame: Day 0 and Day 28 post immunogenicity dose
Population: All participants who received any investigational product (Q=1385; All FM=927), had post dose HAI antibody measurement at the appropriate time and had no protocol deviation judged to have the potential to interfere with the generation or interpretation of an immune response and were seronegative to the strain (Q=364; All FM=244).
Measure: Number; unit: Percent of participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist Group
Number analyzed (Participants) | 364 | 244
Percent of participants | 9.9 | 11.1

12. Secondary Outcome: Percent of Seronegative Participants Within Each Treatment Arm Who Experienced a Seroresponse to the B/Yamagata Strain Post Immunogenicity Dose
Description: as for outcome 10
Time Frame: Day 0 and Day 28 post immunogenicity dose
Population: All participants who received any investigational product (Q=1385; FY=464), had post dose HAI antibody measurement at the appropriate time, had no protocol deviation judged to have the potential to interfere with the generation or interpretation of an immune response, and were seronegative to the strain (Q=483; FY=165).
Measure: Number; unit: Percent of participants
Arm/Group | Q/LAIV (MEDI3250) | FluMist/B/Yamagata
Number analyzed (Participants) | 483 | 165
Percent of participants | 83.0 | 84.8

13. Secondary Outcome: Percent of Seronegative Participants Within Each Treatment Arm Who Experienced a Seroresponse to the B/Victoria Strain Post Immunogenicity Dose
Description: as for outcome 10
Time Frame: Day 0 and Day 28 post immunogenicity dose
Population: All participants who received any investigational product (Q=1385; FV=463), had post dose HAI antibody measurement at the appropriate time, had no protocol deviation judged to have the potential to interfere with the generation or interpretation of an immune response, and were seronegative to the strain (Q=487; FV=159).
Measure: Number; unit: Percent of participants
Arm/Group | Q/LAIV (MEDI3250) | FluMist/B/Victoria
Number analyzed (Participants) | 487 | 159
Percent of participants | 68.8 | 73.6

14. Secondary Outcome: Percent of Participants (Regardless of Serostatus) Who Achieved an A/H1N1 or A/H3N2 Strain-specific HAI Antibody Titer ≥ 32 Post Immunogenicity Dose
Time Frame: Day 28 post immunogenicity dose
Population: All participants who received any investigational product (Q=1385; All FM=927), had post dose HAI antibody measurement at the appropriate time, and had no protocol deviation judged to have the potential to interfere with the generation or interpretation of an immune response (Q=1327; All FM=883).
Measure: Number; unit: Percent of participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist Group
Number analyzed (Participants) | 1327 | 883
Percent of participants
  A/H1N1 | 43.1 | 43.8
  A/H3N2 | 55.7 | 55.4

15. Secondary Outcome: Percent of Participants (Regardless of Serostatus) Who Achieved a B/Yamagata HAI Antibody Titer ≥ 32 Post Immunogenicity Dose
Time Frame: Day 28 post immunogenicity dose
Population: All participants who received any investigational product (Q=1385; FY=464), had post dose HAI antibody measurement at the appropriate time, and had no protocol deviation judged to have the potential to interfere with the generation or interpretation of an immune response (Q=1327; FY=445).
Measure: Number; unit: Percent of participants
Arm/Group | Q/LAIV (MEDI3250) | FluMist/B/Yamagata
Number analyzed (Participants) | 1327 | 445
Percent of participants | 76.5 | 81.6

16. Secondary Outcome: Percent of Participants (Regardless of Serostatus) Who Achieved a B/Victoria HAI Antibody Titer ≥ 32 Post Immunogenicity Dose
Time Frame: Day 28 post immunogenicity dose
Population: All participants who received any investigational product (Q=1385; FV=463), had post dose HAI antibody measurement at the appropriate time, and had no protocol deviation judged to have the potential to interfere with the generation or interpretation of an immune response (Q=1327; FV=437).
Measure: Number; unit: Percent of participants
Arm/Group | Q/LAIV (MEDI3250) | FluMist/B/Victoria
Number analyzed (Participants) | 1327 | 437
Percent of participants | 65.6 | 66.6

17. Secondary Outcome: Percent of Serosusceptible Participants Who Achieved an A/H1N1 HAI Antibody Titer ≥ 32 Post Immunogenicity Dose
Description: Serosusceptible was defined as a baseline HAI titer ≤ 8.
Time Frame: Day 28 post immunogenicity dose
Population: as for outcome 6
Measure: Number; unit: Percent of participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist Group
Number analyzed (Participants) | 569 | 392
Percent of participants | 5.1 | 6.1

18. Secondary Outcome: Percent of Serosusceptible Participants Who Achieved an A/H3N2 HAI Antibody Titer ≥ 32 Post Immunogenicity Dose
Description: Serosusceptible was defined as a baseline HAI titer ≤ 8.
Time Frame: Day 28 post immunogenicity dose
Population: as for outcome 7
Measure: Number; unit: Percent of participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist Group
Number analyzed (Participants) | 435 | 298
Percent of participants | 4.8 | 4.4

19. Secondary Outcome: Percent of Serosusceptible Participants Who Achieved a B/Yamagata HAI Antibody Titer ≥ 32 Post Immunogenicity Dose
Description: Serosusceptible was defined as a baseline HAI titer ≤ 8.
Time Frame: Day 28 post immunogenicity dose
Population: as for outcome 8
Measure: Number; unit: Percent of participants
Arm/Group | Q/LAIV (MEDI3250) | FluMist/B/Yamagata
Number analyzed (Participants) | 588 | 192
Percent of participants | 60.9 | 69.3

20. Secondary Outcome: Percent of Serosusceptible Participants Who Achieved a B/Victoria HAI Antibody Titer ≥ 32 Post Immunogenicity Dose
Description: Serosusceptible was defined as a baseline HAI titer ≤ 8.
Time Frame: Day 28 post immunogenicity dose
Population: as for outcome 9
Measure: Number; unit: Percent of participants
Arm/Group | Q/LAIV (MEDI3250) | FluMist/B/Victoria
Number analyzed (Participants) | 620 | 191
Percent of participants | 41.1 | 44.0

21. Secondary Outcome: Percent of Seronegative Participants Who Achieved an A/H1N1 HAI Antibody Titer ≥ 32 Post Immunogenicity Dose
Description: Seronegative was defined as a baseline HAI titer ≤ 4.
Time Frame: Day 28 post immunogenicity dose
Population: All participants who received any investigational product (Q=1385; All FM=927), had post dose HAI antibody measurement at the appropriate time, had no protocol deviation judged to have the potential to interfere with the generation or interpretation of an immune response, and were seronegative to the strain (Q=460; All FM=321).
Measure: Number; unit: Percent of participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist Group
Number analyzed (Participants) | 460 | 321
Percent of participants | 5.2 | 5.6

22. Secondary Outcome: Percent of Seronegative Participants Who Achieved an A/H3N2 HAI Antibody Titer ≥ 32 Post Immunogenicity Dose
Description: Seronegative was defined as a baseline HAI titer ≤ 4.
Time Frame: Day 28 post immunogenicity dose
Population: All participants who received any investigational product (Q=1385; All FM=927), had post dose HAI antibody measurement at the appropriate time, had no protocol deviation judged to have the potential to interfere with the generation or interpretation of an immune response, and were seronegative to the strain (Q=364; All FM=244).
Measure: Number; unit: Percent of participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist Group
Number analyzed (Participants) | 364 | 244
Percent of participants | 3.8 | 4.9

23. Secondary Outcome: Percent of Seronegative Participants Who Achieved a B/Yamagata HAI Antibody Titer ≥ 32 Post Immunogenicity Dose
Description: Seronegative was defined as a baseline HAI titer ≤ 4.
Time Frame: Day 28 post immunogenicity dose
Population: as for outcome 12
Measure: Number; unit: Percent of participants
Arm/Group | Q/LAIV (MEDI3250) | FluMist/B/Yamagata
Number analyzed (Participants) | 483 | 165
Percent of participants | 60.9 | 70.9

24. Secondary Outcome: Percent of Seronegative Participants Who Achieved a B/Victoria HAI Antibody Titer ≥ 32 Post Immunogenicity Dose
Description: Seronegative was defined as a baseline HAI titer ≤ 4.
Time Frame: Day 28 post immunogenicity dose
Population: All participants who received any investigational product (Q=1385; FY=464), had post dose HAI antibody measurement at the appropriate time, had no protocol deviation judged to have the potential to interfere with the generation or interpretation of an immune response, and were seronegative to the strain (Q=487; FV=159).
Measure: Number; unit: Percent of Participants
Arm/Group | Q/LAIV (MEDI3250) | FluMist/B/Victoria
Number analyzed (Participants) | 487 | 159
Percent of Participants | 37.0 | 42.8

25. Secondary Outcome: Percent of All Participants Experiencing Each Solicited Symptom From Administration of Investigational Product Through 14 Days Post Dose 1
Description: Solicited symptoms were fever ≥ 100.4°F (38.0°C), runny/stuffy nose, sore throat, cough, headache, generalized muscle aches, decreased activity level (lethargy) OR tiredness/weakness, decreased appetite. Collection of specific solicited symptoms (sore throat, headache, generalized muscle aches) was omitted when, according to the judgment of the investigator, the subject was too young to reliably report a particular symptom.
Time Frame: Days 0-14 Post Dose 1
Population: All participants who received any investigational product (Q=1385; All FM=927) and for whom any follow-up solicited symptom safety data were recorded during the summarized period (Q=1377; All FM=920).
Measure: Number; unit: Percent of Participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist Group
Number analyzed (Participants) | 1377 | 920
Percent of Participants
  Any solicited symptom | 47.9 | 47.4
  Fever ≥ 100.4°F (38.0°C) | 5.7 | 3.9
  Fever ≥ 101.3°F (38.5°C) | 3.3 | 2.3
  Fever ≥ 102.2°F (39.0°C) | 1.4 | 0.8
  Fever ≥ 103.1°F (39.5°C) | 0.3 | 0.2
  Fever ≥ 104.0°F (40.0°C) | 0.1 | 0.0
  Fever ≥ 104.9°F (40.5°C) | 0.0 | 0.0
  Runny/stuffy nose | 32.3 | 32.0
  Sore throat | 9.2 | 10.3
  Cough | 15.8 | 16.8
  Headache | 12.5 | 12.2
  Generalized muscle aches | 4.4 | 4.6
  Decreased activity level or tiredness/weakness | 9.8 | 9.9
  Decreased appetite | 5.5 | 6.6

26. Secondary Outcome: Percent of Two-dose Participants Experiencing Each Solicited Symptom From Administration of Investigational Product Through 14 Days Post Dose 1
Description: as for outcome 25
Time Frame: Days 0-14 Post Dose 1
Population: All two-dose participants who received any investigational product (Q=1083; All FM=719) and for whom any follow-up solicited symptom safety data were recorded during the summarized period (Q=1078; All FM=716).
Measure: Number; unit: Percent of Participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist Group
Number analyzed (Participants) | 1078 | 716
Percent of Participants
  Any solicited symptom | 48.1 | 47.5
  Fever ≥ 100.4°F (38.0°C) | 6.6 | 4.2
  Fever ≥ 101.3°F (38.5°C) | 4.0 | 2.2
  Fever ≥ 102.2°F (39.0°C) | 1.7 | 0.8
  Fever ≥ 103.1°F (39.5°C) | 0.4 | 0.3
  Fever ≥ 104.0°F (40.0°C) | 0.1 | 0.0
  Fever ≥ 104.9°F (40.5°C) | 0.0 | 0.0
  Runny/stuffy nose | 33.8 | 31.7
  Sore throat | 8.2 | 8.9
  Cough | 17.2 | 18.0
  Headache | 9.7 | 10.1
  Generalized muscle aches | 4.5 | 4.3
  Decreased activity level or tiredness/weakness | 9.3 | 8.2
  Decreased appetite | 5.6 | 6.7

27. Secondary Outcome: Percent of Two-dose Participants Experiencing Each Solicited Symptom From Administration of Dose 2 During Days 0-14 Post Dose 2
Description: as for outcome 25
Time Frame: Days 0-14 Post Dose 2
Population: All two-dose participants who received any investigational product (Q=1083; All FM=719) and for whom any follow-up solicited symptom safety data were recorded during the summarized period (Q=1039; All FM=692).
Measure: Number; unit: Percent of Participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist Group
Number analyzed (Participants) | 1039 | 692
Percent of Participants
  Any solicited symptom | 31.4 | 30.6
  Fever ≥ 100.4°F (38.0°C) | 2.7 | 4.2
  Fever ≥ 101.3°F (38.5°C) | 1.5 | 2.3
  Fever ≥ 102.2°F (39.0°C) | 0.8 | 1.0
  Fever ≥ 103.1°F (39.5°C) | 0.3 | 0.3
  Fever ≥ 104.0°F (40.0°C) | 0.0 | 0.1
  Fever ≥ 104.9°F (40.5°C) | 0.0 | 0.0
  Runny/stuffy nose | 20.9 | 19.5
  Sore throat | 4.1 | 4.6
  Cough | 12.7 | 11.7
  Headache | 5.4 | 5.5
  Generalized muscle aches | 1.2 | 0.9
  Decreased activity level or tiredness/weakness | 5.9 | 5.3
  Decreased appetite | 3.7 | 3.3

28. Secondary Outcome: Percent of All Participants Experiencing Any Adverse Event From Administration of Investigational Product Through Day 28 Post Dose 1
Description: Any untoward medical occurrence in a patient or clinical investigation in a subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Days 0-28 Post Dose 1
Population: All participants who received any investigational product (Q=1385; All FM=927) and for whom any safety data were recorded during the summarized period (Q=1382; All FM=923).
Measure: Number; unit: Percent of Participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist Group
Number analyzed (Participants) | 1382 | 923
Percent of Participants | 21.0 | 20.7

29. Secondary Outcome: Percent of Two-dose Participants Experiencing Any Adverse Event From Administration of Investigational Product Through Day 28 Post Dose 1
Description: as for outcome 28
Time Frame: Days 0-28 Post Dose 1
Population: All two-dose participants who received any investigational product (Q=1083; All FM=719) and for whom any safety data were recorded during the summarized period (Q=1083; All FM=719).
Measure: Number; unit: Percent of Participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist Group
Number analyzed (Participants) | 1083 | 719
Percent of Participants | 20.3 | 22.9

30. Secondary Outcome: Percent of Two-dose Participants Experiencing Any Adverse Event From Administration of Dose 2 Through 28 Days Post Dose 2
Description: as for outcome 28
Time Frame: Days 0-28 Post Dose 2
Population: All two-dose participants who received any investigational product (Q=1083; All FM=719) and for whom any post Dose 2 safety data were recorded during the summariezed period (Q=1041; All FM=693).
Measure: Number; unit: Percent of participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist Group
Number analyzed (Participants) | 1041 | 693
Percent of participants | 13.4 | 16.7

31. Secondary Outcome: Percent of All Participants Reporting Any Serious Adverse Event (SAE) From Administration of Investigational Product Through Day 28 Post Dose 1
Description: SAEs were those AEs that resulted in death; were immediately life threatening; resulted in inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability or incapacity; were a congenital anomaly in the offspring of a participant; or were an important medical event that may not have resulted in death, threatened life, or required hospitalization and that, based on appropriate medical judgement, may have jeopardized the participant and may have required medical or surgical intervention to prevent on the outcomes listed above.
Time Frame: Days 0-28 Post Dose 1
Population: as for outcome 28
Measure: Number; unit: Percent of participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist Group
Number analyzed (Participants) | 1382 | 923
Percent of participants | 0.0 | 0.0

32. Secondary Outcome: Percent of Two-dose Participants Reporting Any SAE From Administration of Dose 2 During Days 0-28 Post Dose 2
Description: as for outcome 31
Time Frame: Days 0-28 Post Dose 2
Population: All two-dose participants who received any investigational product (Q=1083; All FM=719) and for whom any post Dose 2 safety data were recorded during the summarized period (Q=1041; All FM=693).
Measure: Number; unit: Percent of participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist Group
Number analyzed (Participants) | 1041 | 693
Percent of participants | 0.2 | 0.1

33. Secondary Outcome: Percent of All Participants Reporting Any SAE From Administration of Investigational Product Through 180 Days Post Last Dose
Description: as for outcome 31
Time Frame: Days 0-180 Post Last Dose
Population: as for outcome 28
Measure: Number; unit: Percent of participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist Group
Number analyzed (Participants) | 1382 | 923
Percent of participants | 0.4 | 0.5

34. Secondary Outcome: Percent of All Participants Reporting Any New Onset Chronic Disease (NOCD) From Administration of Investigational Product Through 180 Days Post Last Dose
Description: An NOCD was a newly diagnosed medical condition that was of a chronic, ongoing nature and was assessed by the investigator as medically significant.
Time Frame: Days 0-180 Post Last Dose
Population: as for outcome 28
Measure: Number; unit: Percent of participants
Arm/Group | Q/LAIV (MEDI3250) | All FluMist Group
Number analyzed (Participants) | 1382 | 923
Percent of participants | 1.4 | 0.8

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Day 0 through 28 after Doses 1 and 2. Serious adverse events were collected between Days 0-180 after the last dose administered.
Arm/Group | Q/LAIV (MEDI3250) | All FluMist Group
Serious Adverse Events (participants affected / at risk) | 6/1382 | 5/923
Other Adverse Events (participants affected / at risk) | 176/1382 | 105/923
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Q/LAIV (MEDI3250) (N=1382) | All FluMist Group (N=923)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lung injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Q/LAIV (MEDI3250) (N=1382) | All FluMist Group (N=923)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 10 (12) | 12 (14)
DIARRHOEA (Gastrointestinal disorders) | 22 (22) | 19 (19)
VOMITING (Gastrointestinal disorders) | 36 (37) | 20 (21)
PYREXIA (General disorders) | 23 (23) | 6 (8)
OTITIS MEDIA (Infections and infestations) | 12 (12) | 12 (12)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 8 (8) | 11 (11)
COUGH (Respiratory, thoracic and mediastinal disorders) | 27 (27) | 16 (17)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 22 (23) | 17 (17)
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 16 (17) | 8 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.